CLINICAL TRIAL: NCT05340335
Title: Determination of the Effective Dose 90 of Remimazolam Loading Dose for Adequate Sedation in Patients Undergoing Orthopaedic Surgery Under Monitored Anesthetic Care
Brief Title: ED90 of Remimazolam Loading Dose for Sedation in Patients Under Monitored Anesthetic Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021-2407-0002
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Remimazolam; Orthopedic Procedures; Sedatives
Keywords: remimazolam, sedative effect
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remimazolam (Experimental): A loading dose of remimazolam is administered for sedation
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — A beginning dose of remimazolam is 1mg/kg/hr. When sedation is not achieved in 10 minutes, the dose will be increased by 0.1mg/kg/hr in the next patient. When sedation is successful, the same dose will be used with the probability of 0.89, or the dose will be decreased by 0.1mg/kg/hr with the probability of 0.11 in the next patient. (maximal dose: 2mg/kg/hr)

SUMMARY:
Currently used drugs for monitored general anesthesia include propofol, midazolam, and dexmedetomidine. Each drug has different advantages and disadvantages. Remimazolam causes a relatively small decrease in blood pressure, and it has no injection pain. In addition, remimazolam has a very short onset time, and even after the continuous infusion, the onset of remimazolam is fast, and even after continuous injection, the effect disappeared very quickly due to the short context-sensitive half time. nd through continuous infusion, the patient's depth of anesthesia can be maintained constant. In addition, the short duration of action and the ability to quickly reverse the effect of flumazenil suggest that remimazolam can be used effectively under general anesthesia as well as under general anesthesia. Remimazolam can be used as a continuous infusion for general anesthesia. However, it has also been reported to be used for sedation by continuous infusion or divided intravenous infusion. However, the effective infusion dose of remimazolam for supervised general anesthesia without mechanical ventilation has not been established.

In this study, the ED90 of the loading dose to induce loss of consciousness in patients when supervised general anesthesia is performed through continuous infusion of Remimazolam is to be obtained.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3
* Patients who are scheduled to undergo upper/lower limb surgery under the monitored anesthetic care with remimazolam

Exclusion Criteria:

* Patients who refuse to participate in this study
* Patients with hypersensitivity to benzodiazepine or flumazenil
* Patients with severe renal/hepatic disease
* Patients with drug/alcohol abuse
* Patients who take antidepressants, anticonvulsants, psychoactive drugs chronically
* Patients with difficulty in communication
* Patients with severe obstructive sleep apnea or other airway problems
* Patients contraindicated to regional anesthesia
* Patients judged to be inappropriate for this study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Whether sedation was successful | for 10 minutes from the initiation of the remimazolam administration
  MOAA/S score of 3 or less (MOAA/S: Modified Observer's Alertness/Sedation scale) Awake (5) - Unresponsive (0)

SECONDARY OUTCOMES:
Total amount of remimazolam for sedation | From the initiation of the remimazolam administration to the time when MOAA/S score of 3 or less, assessed up to 10 minutes
  MOAA/S score of 3 or less
Effect site concentration | From the initiation of the remimazolam administration to the time when MOAA/S score of 3 or less, assessed up to 10 minutes
  Calculated by a computerized program(Asanpump)

CONTACTS AND LOCATIONS:
Overall Officials: Ha-Jung Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Kim H, Park HS, Kim HJ, Ro YJ, Koh WU. Effective remimazolam loading dose for adequate sedation in regional anesthesia. Can J Anaesth. 2024 Jun;71(6):818-825. doi: 10.1007/s12630-024-02698-1. Epub 2024 Feb 20. PMID 38378937